CLINICAL TRIAL: NCT07074223
Title: Deep Fascial Graft Versus Acellular Dermal Matrix Conduit on Repaired Hand's Flexor Tendon: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Osama Hassan Elbanna, lecturer of plastic surgery, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tendon fascial graft
Record Dates: First submitted 2025-06-28; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Tendon Injury - Hand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Placebo Comparator): Modefied kestler tendon repair
  Interventions: Procedure: Modified Kestler tendon repair
- Pelnac Group (Experimental): Modified kestler tendon repair wrapped by Pelnac
  Interventions: Procedure: ADM (Pelnac) wrapping of repaired tendon
- Fascia Group (Experimental): modefied kestler tendon repair wrapped by fascial graft
  Interventions: Procedure: Fascial wrapping the site of tendon repair

INTERVENTIONS:
Procedure: Fascial wrapping the site of tendon repair — wrapping the tendon repair site by Pelnac or Fascial graft
  Arms: Fascia Group
Procedure: Modified Kestler tendon repair — Modified Kestler tendon repair
  Arms: Control Group
Procedure: ADM (Pelnac) wrapping of repaired tendon — Modifed kestler tendon repair wrapped by ADM ( Pelnac)
  Arms: Pelnac Group

SUMMARY:
The investigators aim to evaluate the efficacy & applicability of using deep fascial grafts and acellular dermal matrix conduits in reducing post flexor tendon repair adhesions and improving the clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* recent hand cut tendon

Exclusion Criteria:

1. All patients less than 16 years old.
2. Zone 1 , 3 , 4 and zone 5 flexor tendon injuries.
3. Patients with flexor pollicis longus tendon injury.
4. Severely lacerated or crushed tendons.
5. Tendon defects.
6. Multiple level tendon injuries.
7. Associated injuries to muscles.
8. Associated hand or forearm fractures.
9. Patients with poor general condition.
10. Patients with limited passive hand movements.
11. Soft tissues defects overlying the repaired tendons.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participant with treatment related limitation of Movement | 6 months postoperative
  Buck-Gramcko II criteria
Number of participant who have fibrous adhesions in Ultra sonography | 6 months poostoperative
  muscloskeletal ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospitals, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No